CLINICAL TRIAL: NCT01879540
Title: A Phase II, Open-Label, Single-Arm, Multicenter Study to Evaluate the Safety and Immunogenicity of a Trivalent, Surface Antigen Inactivated Subunit Influenza Virus Vaccine Including MF59C.1 Adjuvant (Fluad®) in Healthy Adults ≥65 Years of Age
Brief Title: Safety and Immunogenicity of a Subunit Trivalent Influenza Vaccine, Northern Hemisphere Formulation 2013/2014, Including MF59C.1 Adjuvant, in Healthy Adults ≥65 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70_44S; 2013-000607-16 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Human Influenza
Keywords: Influenza,; Elderly,; Immunology,; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aTIV (Experimental): Adult subjects ≥65 years of age received one dose of a trivalent, surface antigen, inactivated influenza vaccine including MF59C.1 adjuvant (aTIV), formulation 2013/2014 Northern Hemisphere
  Interventions: Biological: aTIV

INTERVENTIONS:
Biological: aTIV — Adjuvanted Trivalent Influenza Virus Vaccine (surface antigen, inactivated, adjuvanted with MF59C.1, egg-derived)

SUMMARY:
The present study is designed to confirm the safety and immunogenicity of trivalent, surface antigen, inactivated influenza vaccine including MF59C.1 adjuvant, formulation 2013/2014 Northern Hemisphere, in adults ≥65 years of age.

For the immunogenicity endpoints the antibody response to each influenza vaccine antigen, will be measured by means of Single Radial Hemolysis (SRH) or Hemagglutination Inhibition (HI) at approximately 21 days post immunization.

The vaccine composition will be based on the World Health Organization (WHO) recommended influenza strains for 2013/2014 Northern Hemisphere.

The results of this study are intended to support the use of this vaccine in future influenza seasons if the recommended vaccine composition remains the same, in compliance with the requirements of the current European Union (EU) recommendations for clinical trials related to yearly licensing of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged 65 years or older, mentally competent, who gave written informed consent prior to study entry;
* Were able to comply with all the study requirements; and
* Were in good health as determined by the outcome of medical history, physical examination, and clinical judgment of the investigator.

Exclusion Criteria:

* Had behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may have interfered with the subject's ability to participate in the study;
* Had a serious chronic or acute disease (in the judgment of the investigator) including, but not limited to:

  * medically significant cancer (except for benign or localized skin cancer, cancer in remission for >= 10 years, or localized prostate cancer that has been clinically stable for > 2 years without treatment)
  * medically significant advanced congestive heart failure (ie, New York Heart Association [NYHA] class III and IV)
  * chronic obstructive pulmonary disease (ie, Global initiative for chronic Obstructive Lung Disease [GOLD] stage III and IV)
  * autoimmune disease (including rheumatoid arthritis and excepting Hashimoto's thyroiditis that has been clinically stable for >= 5 years)
  * diabetes mellitus type I
  * poorly controlled diabetes mellitus type II
  * advanced arteriosclerotic disease
  * history of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (eg, Down's syndrome)
  * acute or progressive hepatic disease
  * acute or progressive renal disease
  * severe neurological (especially Guillain-Barré syndrome) or psychiatric disorder
  * severe asthma
* Had a history of any anaphylactic reaction and/or serious allergic reaction to any component of the study vaccine.
* Had a known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:

  * receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study,
  * receipt of immunostimulants within the past 6 months,
  * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within the past 3 months and for the full length of the study, or
  * suspected or known human immunodeficiency virus (HIV) infection or HIV related disease.
* Had known or suspected drug or alcohol abuse within the past 2 years;
* Had bleeding diathesis or conditions associated with prolonged bleeding time that, in the investigator's opinion, would have interfered with the safety of the subject;
* Was not able to comprehend and to follow all required study procedures for the whole period of the study;
* Had a history or any illness that, in the opinion of the investigator, would have posed additional risk to the subjects because of participation in the study;
* Had the following within the past 6 months:

  * any laboratory confirmed seasonal or pandemic influenza disease,
  * received any seasonal or pandemic influenza vaccine.
* Had received any other vaccine within 4 weeks prior to enrollment in this study or who were planning to receive any vaccine during the study;
* Had acute or chronic infections requiring antiviral therapy within the last 7 days;
* Had experienced fever (ie, body temperature [preferably oral] >= 38.0°C) within the last 3 days of intended study vaccination;
* Had been participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intended to participate in another clinical study at any time during the conduct of this study;
* Was part of study personnel or had close family members conducting this study;
* Had a body mass index (BMI) >35 kg/m2 (BMI is calculated by dividing the subject's weight in kilograms by the subject's height in meters multiplied by the subject's height in meters)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (1):
- Antwerp University Centre for the Evaluation of Vaccination, Antwerp, Wilrijk, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | aTIV
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | aTIV
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: year] | 71.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Single Radial Hemolysis (SRH) Areas ≥25mm2, Against Each of Three Vaccine Strains After Receiving One Dose of aTIV
Description: Immunogenicity was assessed in terms of percentages of adult subjects ≥65 years of age with SRH areas ≥25mm2 against each of the three vaccine strains, three weeks after receiving one dose of aTIV.
  The related European Committee for Human Medicinal Products (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving post vaccination SRH areas ≥ 25mm2 is >60%.
Time Frame: Day 1 (baseline) and Day 22
Population: Analysis was done on the per-protocol population i.e all subjects who have received study vaccination and provided immunogenicity data both at baseline and after vaccination; did not withdraw informed consent and did not have Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) confirmed influenza during the study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV
Number analyzed (Participants) | 61
Percentage of subjects
  Day 1 (H1N1 strain) | 46 [33 to 59]
  Day 22 (H1N1 strain) | 89 [78 to 95]
  Day 1 (H3N2 strain) | 43 [30 to 56]
  Day 22 (H3N2 strain) | 90 [80 to 96]
  Day 1 (B strain) | 28 [17 to 41]
  Day 22 (B strain) | 79 [66 to 88]

2. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in SRH Area, Against Each of Three Vaccine Strains After Receiving One Dose of aTIV
Description: Immunogenicity was assessed in terms of percentages of adult subjects ≥65 years of age achieving seroconversion or significant increase in SRH area against each of the three vaccine strains, three weeks after receiving one dose of aTIV.
  Seroconversion is defined as percentage of subjects with a pre-vaccination SRH area ≤4mm2 achieving a post-vaccination SRH area ≥25 mm2. Significant increase is defined as percentage of subjects with a pre-vaccination SRH area >4mm2 achieving at least 50% increase in post-vaccination SRH area.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if>30% of subjects achieve seroconversion or significant increase in post-vaccination SRH area.
Time Frame: Day 22
Population: Analysis was done on the per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV
Number analyzed (Participants) | 61
Percentage of subjects
  H1N1 strain | 57 [44 to 70]
  H3N2 strain | 61 [47 to 73]
  B strain | 70 [57 to 81]

3. Primary Outcome: Geometric Mean Ratio (GMR) of Post Vaccination Versus Pre Vaccination Geometric Mean Areas (GMAs), Against Each of Three Vaccine Strains After Receiving One Dose of aTIV
Description: The antibody responses following one dose of aTIV were evaluated in terms of geometric mean ratio GMRs of post vaccination GMAs to pre vaccination GMAs against each of the three vaccine strains, three weeks after receiving one dose of aTIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is > 2.0.
Time Frame: Day 22/Day 1
Population: Analysis was done on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | aTIV
Number analyzed (Participants) | 61
Ratio
  H1N1 strain | 2.63 [2.04 to 3.39]
  H3N2 strain | 2.34 [1.91 to 2.87]
  B strain | 2.89 [2.35 to 3.57]

4. Primary Outcome: Percentages of Subjects With Haemagglutinin Inhibition(HI) Titers ≥40, Against Each of Three Vaccine Strains After Receiving One Dose of aTIV.
Description: Immunogenicity was assessed in terms of percentages of adult subjects ≥65 years of age with HI titers ≥40, against each of the three vaccine strains, three weeks after receiving one dose of aTIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the of subjects achieving HI titers ≥ 40 is >60%.
Time Frame: Day 1 (baseline) and Day 22
Population: Analysis was done on the per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV
Number analyzed (Participants) | 61
Percentage of subjects
  Day 1 (H1N1 strain) | 75 [63 to 86]
  Day 22 (H1N1 strain) | 97 [89 to 100]
  Day 1 (H3N2 strain) | 89 [78 to 95]
  Day 22 (H3N2 strain) | 100 [94 to 100]
  Day 1 (B strain) | 61 [47 to 73]
  Day 22 (B strain) | 98 [91 to 100]

5. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in HI Antibody Titers, Against Each of Three Vaccine Strains After Receiving One Dose of aTIV
Description: Immunogenicity was assessed in terms of percentages of adult subjects ≥65 years of age achieving seroconversion or significant increase in HI antibody titers after receiving one dose of aTIV.
  Seroconversion is defined as percentage of subjects with a pre-vaccination HI titer <10 to a post-vaccination titer ≥40. Significant increase is defined as percentage of subjects with a pre-vaccination HI titer ≥10 to at least a 4-fold increase in post-vaccination HI antibody titers.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if >30% of subjects achieve seroconversion or significant increase in post-vaccination HI titers.
Time Frame: Day 22
Population: Analysis was done on the per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV
Number analyzed (Participants) | 61
Percentage of subjects
  H1N1 strain | 39 [27 to 53]
  H3N2 strain | 43 [30 to 56]
  B strain | 38 [26 to 51]

6. Primary Outcome: Geometric Mean Ratio (GMR) of Post Vaccination Versus Pre Vaccination HI Titers, Against Each of Three Vaccine Strains After Receiving One Dose of aTIV
Description: The antibody responses following one dose of aTIV were evaluated in terms of GMRs of post vaccination geometric mean HI titers against each of the three vaccine strains, three weeks after receiving one dose of aTIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is > 2.0.
Time Frame: Day 22/Day 1
Population: Analysis was done on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | aTIV
Number analyzed (Participants) | 61
Ratio
  H1N1 strain | 3.57 [2.59 to 4.91]
  H3N2 strain | 3.32 [2.45 to 4.49]
  B strain | 2.69 [2.22 to 3.26]

7. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events After Receiving One Dose of aTIV
Description: The number of adult subjects ≥65 years of age reporting solicited local and systemic adverse events and other solicited adverse events after receiving one dose of aTIV are reported.
Time Frame: Day 1 to Day 4 post vaccination
Population: Analysis was done on the safety set population i.e all subjects who have post-vaccination AE or reactogenicity records
Measure: Number; unit: Participants
Arm/Group | aTIV
Number analyzed (Participants) | 63
Participants
  Any Local | 26
  Injection site induration | 2
  Injection site erythema | 3
  Injection site ecchymosis | 2
  Injection site pain | 21
  Any systemic | 15
  Chills/shivering | 1
  Malaise | 2
  Myalgia | 2
  Arthralgia | 1
  Fatigue | 11
  Headache | 5
  Fever (≥ 38°C) | 0
  Temperature ≥40°C | 0
  Prophylactic use of analgesics/antipyretics (N=61) | 0
  Therapeutic use of analgesics/antipyretics (N=61) | 2

8. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving One Dose of aTIV
Description: The number of adult subjects ≥65 years of age subjects reporting any unsolicited adverse event (AEs) between Day 1 to 4 and serious adverse events (SAEs), medically attended AEs, AEs leading to withdrawal from the study between Day 1 to Day 22 after receiving one dose of aTIV are reported.
Time Frame: Day 1 to Day 22 post-vaccination
Population: Analysis was done on the unsolicited safety set population i.e all subjects who had post-vaccination unsolicited AE records
Measure: Number; unit: Participants
Arm/Group | aTIV
Number analyzed (Participants) | 63
Participants
  Any AE | 12
  At least possibly related AEs | 10
  Serious AEs | 0
  At least possibly related SAEs | 0
  Medically attended AEs | 5
  AEs leading to withdrawal | 0
  Death | 0

ADVERSE EVENTS:
Time Frame: All solicited AEs and unsolicited AEs were collected from Day 1 to Day 4; all unsolicited SAEs, medically attended AEs, AEs leading to withdrawal from the study were collected from Day 1 to Day 22
Arm/Group | aTIV
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 32/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aTIV (N=63)
Fatigue (General disorders) | 11
Injection site erythema (General disorders) | 5
Injection site pain (General disorders) | 21
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less